CLINICAL TRIAL: NCT02350296
Title: 2-way Crossover, Single Dose Randomized Bioequivalence Phase I Study of Ketoprofen Lysine Salt as Immediate Release Tablets Formulation (40 mg) vs. Oral Solution (80 mg, Half Sachet) After Oral Administration to Healthy Volunteers.
Brief Title: Crossover, Single Dose Randomized, Bioequivalence of Ketoprofen Lysine Salt Immediate Release vs Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KSL0114
Record Dates: First submitted 2014-12-15; First posted 2015-01-29 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pain Disorders
Keywords: headache; dental pain; neuralgia; dysmenorrhoea; muscular and osteoarticular pain
MeSH Terms: conditions — Somatoform Disorders; Headache; Toothache; Neuralgia; Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Reference (KSL 40 mg - OKi® 80 mg) (Experimental): In this arm, a single dose of the test product (1 tablet; 40 mg KLS) was orally administered, under fasting conditions, in the first study period (day 1, 08:00±1h), and, after a wash-out period of at least 4 days, a single dose of the reference product OKi® 80 mg (half a sachet, 40 mg KLS) was orally administered, under fasting conditions, in the second study period (day 1, Visit 5, 08:00 ±1h).
  Interventions: Drug: KSL 40 mg; Drug: OKi® 80 mg
- Reference - Test (OKi® 80 mg - KSL 40 mg) (Experimental): In this arm, a single dose of the reference product OKi® 80 mg (half a sachet, 40 mg KLS) was orally administered, under fasting conditions, in the first study period (day 1, Visit 3, 08:00 ±1h) and, after a wash-out period of at least 4 days, a single dose of the test product (1 tablet; 40 mg KLS) was orally administered, under fasting conditions, in the second study period (day 1, Visit 5, 08:00±1h).
  Interventions: Drug: KSL 40 mg; Drug: OKi® 80 mg

INTERVENTIONS:
Drug: KSL 40 mg — Ketoprofen lysine salt (KLS) immediate release oral tablets 40 mg, corresponding to 25 mg of ketoprofen free acid. Ketoprofen lysine salt was administered according to the randomisation list and the cross-over design. One (1) tablet of test formulation was administered to the subjects in the morning with 240 mL of still mineral water. Afterwards, no fluid intake was permitted for 2 h. All subjects were under fasting conditions from the evening before investigational product administration (i.e. for at least 10 h, overnight).
  Other Names: Ketoprofen lysine salt
Drug: OKi® 80 mg — OKi® 80 mg granules for oral solution (bipartite sachets: each half sachet containing 40 mg of KLS corresponding to 25 mg of ketoprofen free acid). Ketoprofen lysine salt was administered according to the randomisation list and the cross-over design.
  The content of half sachet of the reference formulation was dissolved in 190 mL of still mineral water. The subject drank the entire solution immediately. Then the glass was rinsed with 50 mL of still mineral water and the subject drank the rinse immediately. Afterwards, no fluid intake was permitted for 2 h. All subjects were under fasting conditions from the evening before investigational product administration (i.e. for at least 10 h, overnight).
  Other Names: Ketoprofen lysine salt

SUMMARY:
Objectives:

The objective of the study was to investigate the bioequivalence between two formulations containing ketoprofen lysine salt (KLS) when administered as single oral doses in two consecutive study periods to healthy male and female volunteers under fasting conditions.

Primary end-point: to evaluate the bioequivalent rate (Cmax) and extent (AUC0-t) of absorption of ketoprofen after single dose administration of test and reference products.

Secondary end-points:

* to describe the pharmacokinetic (PK) profile of ketoprofen after single dose administration of test and reference products;
* to collect safety and tolerability data after single dose administration of test and reference products.

DETAILED DESCRIPTION:
This was a single centre, single dose, open, randomised, two-way cross-over, two-stage bioequivalence study. According to the two-stage design of the study, an initial group of subjects was treated in study stage 1 and data were analysed. Since bioequivalence was demonstrated, according to the protocol the study was terminated after stage 1, and stage 2 was not performed.

The study was conducted as planned and consisted of a screening visit, a treatment phase of 2 study periods separated by a wash-out interval of at least 4 days and a final visit / early termination visit (ETV).

Considering the lack of information about the PK profile of the new formulation, it was decided to use a "two stage" bioequivalence study design, that allows a re-calculation of the sample size in case the number of subjects initially enrolled in the study is not large enough to provide a reliable answer to the questions addressed, due to a possible underestimation of the variability or misleading estimation of the point estimate for the test/reference ratio of the geometric means.

The sequence of treatments in the two study periods was assigned to each randomised subject according to a computer generated randomisation list.

A wash-out period of at least 4 days between the two administrations is justified by the elimination half-life of the ketoprofen (1-2 h).

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, subjects must fulfil all these criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: males/females, 18-55 years old inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, pulse rate (PR) 50-90 bpm and body temperature (BT) ≤ 37.5° C, measured after 5 min of rest in the sitting position;
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential and with an active sexual life must be using at least one of the following reliable methods of contraception:

   * Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   * A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   * A male sexual partner who agrees to use a male condom with spermicide
   * A sterile sexual partner

Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, pregnancy test result must be negative at screening.

Exclusion Criteria:

Subjects meeting any of these criteria will not be enrolled in the study:

1. Electrocardiogram (ECG 12-leads, supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principles (ketoprofen) and/or formulations' ingredients; history of hypersensitivity to drugs (in particular to NSAIDs) or allergic reactions in general, which the Investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory (including asthma), skin, haematological, endocrine or neurological and autoimmune diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) drugs [in particular ketoprofen and acetylsalicylic acid (ASA) and NSAIDs in general], herbal remedies and food supplements taken 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study (date of the informed consent signature)
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [> 1 drink/day for females and > 2 drinks/day for males, defined according to the USDA Dietary Guidelines 2010 (6)], caffeine (> 5 cups coffee/tea/day) or tobacco abuse (≥ 6 cigarettes/day)
10. Drug test: positive result at the drug test at screening
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (< 1600 or > 3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2015-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research S.A., Phase I Unit
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 healthy volunteers were randomized, receiving a single dose of Test and Reference treatment. Based on the cross-over design, a single dose of product was given orally in one of the two possible sequences: in the "test-reference" arm, subjects received Ketoprofen lysine salt (KLS) firstly and then the reference product OKI. In the "Reference-Test" arm, subjects received reference product OKi first, then Ketoprofen lysine salt (KLS)"). A wash-out interval separated the 2 treatment periods.
Groups:
- Sequence "Test - Reference": Participants first received a single dose of Ketoprofen lysine salt (KLS, Test product)), 40 mg immediate release tablets (corresponding to 25 mg ketoprofen) under fasting conditions (day 1). After a washout interval of at least 4 days, the participants then received a single dose of the reference product OKi®, KLS 40 mg granules for oral solution, always under fasting conditions (day 1). This according to the study randomised cross-over design.
  There were no premature discontinuations during the study
- Sequence "Reference - Test": Participants first received a single dose of the reference product OKi®, KLS 40 mg granules for oral solution, under fasting conditions (day 1). After a washout interval of at least 4 days, the participants then received a single dose of Ketoprofen lysine salt (KLS, Test product)), 40 mg immediate release tablets (corresponding to 25 mg ketoprofen) always under fasting conditions (day 1).This according to the study randomized cross-over design.
Period: First Treatment Period
Arm/Group | Sequence "Test - Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Washout Period (at Least 4 Days)
Arm/Group | Sequence "Test - Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Treatment Period
Arm/Group | Sequence "Test - Reference" | Sequence "Reference - Test"
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 30 randomised subjects completed the study per protocol and were included in the PK and Safety sets.
Groups:
- All Study Participants: Enrolled Set: all enrolled subjects. This analysis set was used for the analysis of demographic, baseline and background characteristics.
  Safety Set: all subjects who received at least one dose of investigational medicinal product.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 30

OUTCOME MEASURES:

1. Primary Outcome: Ketoprofen Plasma PK Parameters: Cmax
Description: Cmax = maximum plasma concentration. Cmax a of ketoprofen was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentrations of ketoprofen were measured in each study period at the timepoints hereunder reported. Arithmetic means + standard deviation are reported hereunder.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-dose
Population: PK set: all randomised subjects who fulfilled the study protocol requirements in terms of investigational medicinal products intake and have evaluable PK data readouts for the planned treatment comparisons, with no major deviations that could affect the PK results.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- KSL 40 mg (Test Product): Ketoprofen lysine salt (KLS) immediate release tablets 40 mg, corresponding to 25 mg of ketoprofen free acid. A single dose of the test product (1 tablet; 40 mg KLS) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, 08:00±1h), according to the study randomised cross-over design.
  KSL 40 mg: Ketoprofen lysine salt oral immediate release tablets 40 mg. The two single dose administrations (test and reference) in the two study periods were separated by a wash-out interval of at least 4 days.
- OKi® 80 mg (Reference Product): OKi® 80 mg granules for oral solution (bipartite sachets: each half sachet containing 40 mg of KLS corresponding to 25 mg of ketoprofen free acid). A single dose of the reference product (half a sachet, 40 mg KLS) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, 08:00 ±1h), according to the study randomised cross-over design.
  OKi® 80 mg: Ketoprofen lysine salt granules for oral solution 40 mg (half of a bipartite sachet).The two single dose administrations (reference and test) in the two study periods were separated by a wash-out interval of at least 4 days.
Arm/Group | KSL 40 mg (Test Product) | OKi® 80 mg (Reference Product)
Number analyzed (Participants) | 30 | 30
μg/mL | 3.61 (1.17) | 3.40 (1.38)
Statistical Analysis 1: Comparison: KSL 40 mg (Test Product) vs OKi® 80 mg (Reference Product); Test type: Equivalence — Acceptance criterion for bioequivalence was a 94.12% confidence interval for the test/reference ratio of the geometric means within the 80.00-125.00% range, according to the current guidelines for bioequivalence studies; p = 0.1455, ANOVA — "treatment" P value reported; geometric means ratio = 108.12, 94.12% CI 2-sided [97.57 to 119.81] — Estimated value and limits are expressed in %

2. Primary Outcome: Ketoprofen Plasma PK Parameters: AUC0-t
Description: AUC0-t = Area under the concentration-time curve from administration to the last observed concentration time t, calculated with the linear trapezoidal method. AUC0-t of ketoprofen was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentrations of ketoprofen were measured in each study period at the timepoints hereunder specified.
  Please note that AUC0-t was considered a reliable estimate of the extent of absorption if the ratio AUC0-t/AUC0-∞ equalled or exceeded a factor of 0.8, i.e. if %AUCextra was < 20%. Arithmetic means + standard deviation are reported hereunder.
Time Frame: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Groups:
- KSL 40 mg: Ketoprofen lysine salt (KLS) immediate release tablets 40 mg, corresponding to 25 mg of ketoprofen free acid. A single dose of the test product (1 tablet; 40 mg KLS) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, 08:00±1h), according to the study randomised cross-over design.
  KSL 40 mg: Ketoprofen lysine salt oral immediate release tablets 40 mg. The two single dose administrations (test and reference) in the two study periods were separated by a wash-out interval of at least 4 days.
- OKi® 80 mg: OKi® 80 mg granules for oral solution (bipartite sachets: each half sachet containing 40 mg of KLS corresponding to 25 mg of ketoprofen free acid). A single dose of the reference product (half a sachet, 40 mg KLS) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, 08:00 ±1h), according to the study randomised cross-over design.
  OKi® 80 mg: Ketoprofen lysine salt granules for oral solution 40 mg (half of a bipartite sachet).The two single dose administrations (reference and test) in the two study periods were separated by a wash-out interval of at least 4 days.
Arm/Group | KSL 40 mg | OKi® 80 mg
Number analyzed (Participants) | 30 | 30
h*μg/mL | 4.53 (1.35) | 4.12 (1.35)
Statistical Analysis 1: Comparison: KSL 40 mg vs OKi® 80 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0023, ANOVA — "Treatment" P value is reported; geometric means ratio = 110.62, 94.12% CI 2-sided [104.26 to 117.38] — Estimated value and limits are expressed in %

3. Secondary Outcome: Ketoprofen Plasma PK Parameters: AUC0-∞
Description: AUC0-∞ = Area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as AUC0-t + Ct/λz, where Ct is the last measurable drug concentration. AUC0-∞ of ketoprofen was calculated from plasma concentrations after single oral dose of test and reference products. Plasma concentrations of ketoprofen were measured in each study period at the timepoints hereunder reported. Arithmetic means + standard deviation are reported hereunder.
Time Frame: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | KSL 40 mg | OKi® 80 mg
Number analyzed (Participants) | 30 | 30
h*μg/mL | 4.64 (1.40) | 4.22 (1.39)
Statistical Analysis 1: Comparison: KSL 40 mg vs OKi® 80 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0021, ANOVA — "treatment" P value is reported; geometric means ratio = 110.69, 94.12% CI 2-sided [104.35 to 117.41] — Estimated value and limits are expressed in %

4. Secondary Outcome: Ketoprofen Plasma PK Parameters: Tmax
Description: Tmax = Time to achieve Cmax. Tmax (0-8 hours) of ketoprofen calculated from plasma concentrations after single oral dose of test and reference. Plasma concentrations of ketoprofen were measured in each study period at the following timepoints: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose.
Time Frame: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | KSL 40 mg | OKi® 80 mg
Number analyzed (Participants) | 30 | 30
h | 0.39 (0.19) | 0.30 (0.10)
Statistical Analysis 1: Comparison: KSL 40 mg vs OKi® 80 mg; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0201, Friedman

5. Secondary Outcome: Ketoprofen Plasma PK Parameters: T1/2
Description: T1/2 = Half-life, calculated, if feasible, as ln2/λz. T1/2 (0-8 hours) of ketoprofen was calculated from plasma concentrations after single oral dose of test and reference. Plasma concentrations of ketoprofen were measured in each study period at the following timepoints: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose.
Time Frame: pre-dose (0), 5, 15, 30, 45 min, 1, 1.5, 2, 3, 4, 5, 6 and 8 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | KSL 40 mg | OKi® 80 mg
Number analyzed (Participants) | 30 | 30
h | 1.64 (0.17) | 1.64 (0.17)

6. Secondary Outcome: Ketoprofen Plasma PK Parameters: Frel
Description: Frel = Relative bioavailability, calculated as ratio AUC0-t (test)/ AUC0-t (reference)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % of bioavailability
Groups:
- All Participants: Ketoprofen lysine salt (KLS) immediate release tablets 40 mg, corresponding to 25 mg of ketoprofen free acid. A single dose of the test product (1 tablet; 40 mg KLS) was orally administered, under fasting conditions, in one of the two consecutive study periods (day 1, 08:00±1h), according to the study randomised cross-over design.
  KSL 40 mg: Ketoprofen lysine salt oral immediate release tablets 40 mg. The two single dose administrations (test and reference) in the two study periods were separated by a wash-out interval of at least 4 days.
Arm/Group | All Participants
Number analyzed (Participants) | 30
% of bioavailability | 112.07 (18.70)

7. Secondary Outcome: Number of TEAEs
Description: TEAE = Treatment Emergent Adverse Events. TEAEs were assessed throughout the study, from informed consent up to the final visit / early termination visit (ETV), which takes place after visit 5 on day 1 of period 2, more precisely after the 8 h blood sampling and vital signs check.
Time Frame: From Day -14 to Day 1 of period 2 (Final visit/ETV), approximately 1 month
Population: Safety Set: all subjects who received at least one dose of investigational medicinal product.
Measure: Number; unit: number of events
Arm/Group | KSL 40 mg (Test Product) | OKi® 80 mg (Reference Product)
Number analyzed (Participants) | 30 | 30
number of events
  TEAE related to treatment | 1 | 2
  TEAE not related to treatment | 0 | 0
  mild | 1 | 2
  moderate | 0 | 0
  severe | 0 | 0
  TEAE leading to discontinuation | 0 | 0
  serious TEAE | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were assessed throughout the study, from informed consent up to the final visit / early termination visit (ETV), which takes place after visit 5 on day 1 of period 2, more precisely after the 8 h blood sampling and vital signs check. From Day -14 to Day 1 of period 2 (Final visit/ETV), approximately 1 month.
Description: More specifically, adverse events are assessed at:
  Visit 1: days -14/-2 Visit 2: day -1 Visit 3: day 1 Visit 4: Day -1 Visit 5: day 1 From Period 1 to Period 2 : wash-out period of at least 4 days
Arm/Group | KSL 40 mg | OKi® 80 mg
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KSL 40 mg (N=30) | OKi® 80 mg (N=30)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT02350296/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT02350296/SAP_001.pdf